CLINICAL TRIAL: NCT02961790
Title: A Phase III, Double-Blind, Controlled Trial of Oxybutynin in the Management of Hot Flashes
Brief Title: Oxybutynin Chloride in Managing Hot Flashes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ACCRU-SC-1603; NCI-2016-01603 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-SC-1603 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2018-08

CONDITIONS: Breast Carcinoma; Ductal Breast Carcinoma In Situ; Hot Flashes; Lobular Breast Carcinoma In Situ; No Evidence of Disease
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Hot Flashes; Breast Carcinoma In Situ | interventions — oxybutynin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group I (low-dose oxybutynin chloride) (Experimental): Patients receive lower dose oxybutynin chloride PO BID on days 8-49 in the absence of unacceptable toxicity.
  Interventions: Drug: Oxybutynin Chloride; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (low-dose placebo) (Placebo Comparator): Patients receive lower dose placebo PO BID on days 8-49 in the absence of unacceptable toxicity.
  Interventions: Other: Placebo; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group III (high-dose oxybutynin chloride) (Experimental): Patients receive lower dose oxybutynin chloride PO BID on days 8-14 and higher dose oxybutynin chloride on days 15-49 in the absence of unacceptable toxicity.
  Interventions: Drug: Oxybutynin Chloride; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group IV (high-dose placebo) (Placebo Comparator): Patients receive lower dose placebo PO BID on days 8-14 and higher dose placebo on days 15-49 in the absence of unacceptable toxicity.
  Interventions: Other: Placebo; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Oxybutynin Chloride — Given PO
  Other Names: Ditropan; Gelnique; MJ-4309-1; Oxybutynin Hydrochloride
  Arms: Group I (low-dose oxybutynin chloride); Group III (high-dose oxybutynin chloride)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Group II (low-dose placebo); Group IV (high-dose placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase III trial studies how well oxybutynin chloride works in managing hot flashes in patients who are not candidates for, or not interested in hormone replacement therapy. Previous studies have shown that oxybutynin is effective in managing hot flashes, however doses used in prior studies have resulted in side effects. This trial is evaluating lower doses of oxybutynin with the goal of determining if they are efficacious with less side effects.

ADAM-VTE

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether oxybutynin chloride (oxybutynin) can diminish hot-flash activity in women with a history of breast cancer or in women who have a concern about taking estrogen for fear of breast cancer.

SECONDARY OBJECTIVES:

I. To perform a dose-response evaluation of two oxybutynin doses. II. To determine the toxicity of oxybutynin in the study population. III. To assess the impact of hot-flash activity on overall quality of life and to examine whether oxybutynin can diminish this impact on quality of life.

OUTLINE: Patients are randomized into 1 of 4 groups.

GROUP I (LOW-DOSE OXUBUTYNIN CHLORIDE): Patients receive lower dose oxybutynin chloride orally (PO) twice a day (BID) on days 8-49 in the absence of unacceptable toxicity.

GROUP II (LOW-DOSE PLACEBO): Patients receive lower dose placebo PO BID on days 8-49 in the absence of unacceptable toxicity.

GROUP III (HIGH-DOSE OXUBUTYNIN CHLORIDE): Patients receive lower dose oxybutynin chloride PO BID on days 8-14 and higher dose oxybutynin chloride on days 15-49 in the absence of unacceptable toxicity.

GROUP IV (HIGH-DOSE PLACEBO): Patients receive lower dose placebo PO BID on days 8-14 and higher dose placebo on days 15-49 in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* History of breast cancer, ductal breast carcinoma in situ (DCIS), or lobular carcinoma in situ (LCIS) (currently without evidence of malignant disease) OR a concern about taking estrogen for fear of breast cancer
* Bothersome hot flashes (defined by their occurrence of >= 28 times per week and of sufficient severity to prompt the patient to seek therapeutic intervention)
* Presence of hot flashes for > 30 days prior to study entry
* Ability to complete questionnaire(s) by themselves or with assistance
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) = 0, 1
* Ability to provide informed written consent
* Life expectancy >= 6 months
* Willing to work with the enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Any of the following current (=< 4 weeks prior) or planned therapies:

  * Antineoplastic chemotherapy (anti-HER2 agents allowed)
  * Androgens
  * Estrogens (any delivery route)
  * Progestogens
  * Tamoxifen, raloxifene and aromatase inhibitors are allowed, but patient must have been on a constant dose for at least 28 days and must not be expected to stop the medication during the study period
  * Selective serotonin reuptake inhibitors (SSRIs)/serotonin?norepinephrine reuptake inhibitors (SNRIs), when being used for hot flash management or other indications such as depression, is allowed, assuming the dose will remain unchanged for the study duration
  * Gabapentin/pregabalin, when being used for hot flash management (use for other indications, such as pain, is allowed, assuming the dose will remain unchanged for the study duration)
  * Clonidine
  * Agents with known potent anticholinergic activity; agents with mild-moderate anticholinergic activity are allowed
* Prior use of oxybutynin during the period in which patient has had hot flashes
* Pregnant women
* Nursing women
* History of any of the following contraindications to oxybutynin:

  * Uncontrolled gastroesophageal reflux disease (GERD) despite appropriate therapy; if patient has history of GERD, but symptoms are well-controlled with medical treatment, patient is eligible
  * Ulcerative colitis
  * Narrow-angle glaucoma
  * Urinary retention
  * Hypersensitivity to oxybutynin or any other components of the product
  * Current uncontrolled hyperthyroidism
  * Coronary heart disease (angina or prior myocardial infarction)
  * Congestive heart failure
  * Symptomatic cardiac arrhythmias
  * Current uncontrolled hypertension
  * Myasthenia gravis
  * Dementia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, Principal Investigator — Academic and Community Cancer Research United
Locations (13):
- United States (13):
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Carle Cancer Center NCI Community Oncology Research Program, Urbana, Illinois
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Waverly Hematology Oncology, Cary, North Carolina
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Saint Vincent Hospital -Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- High-dose Oxybutynin Chloride Group: Patients receive lower dose oxybutynin chloride PO BID on days 8-14 and higher dose oxybutynin chloride on days 15-49 in the absence of unacceptable toxicity.
- Low-dose Oxybutynin Chloride Group: Patients receive lower dose oxybutynin chloride PO BID on days 8-49 in the absence of unacceptable toxicity.
- High-dose Placebo Group: Patients receive lower dose placebo PO BID on days 8-14 and higher dose placebo on days 15-49 in the absence of unacceptable toxicity.
- Low-dose Placebo Group: Patients receive lower dose placebo PO BID on days 8-49 in the absence of unacceptable toxicity.
Period: Overall Study
Arm/Group | High-dose Oxybutynin Chloride Group | Low-dose Oxybutynin Chloride Group | High-dose Placebo Group | Low-dose Placebo Group
Started | 50 | 51 | 24 | 25
Completed | 35 | 40 | 18 | 20
Not Completed | 15 | 11 | 6 | 5
Not completed — Canceled | 4 | 5 | 1 | 4
Not completed — without baseline data | 4 | 0 | 1 | 0
Not completed — without post baseline data | 7 | 6 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-dose Oxybutynin Chloride Group | Low-dose Oxybutynin Chloride Group | High-dose Placebo Group | Low-dose Placebo Group | Total
Number analyzed (Participants) | 35 | 40 | 18 | 20 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (8.4) | 55.6 (8.0) | 57.5 (8.2) | 58.8 (8.7) | 57.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 40 | 18 | 20 | 113
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 0 | 0 | 3
  White | 34 | 36 | 18 | 20 | 108
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 33 | 36 | 16 | 20 | 105
    1 | 2 | 4 | 2 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Hot Flash Activity Score From Baseline to Week 7 for Low Dose Oxybutynin vs Placebo and for High Dose Oxybutynin vs Placebo
Description: Average change in hot flash activity score from baseline to Week 7 for Low Dose Oxybutynin vs Placebo. The hot flash activity will be measured by the weekly average hot flash score (Sloan JA, et. al., 2001), which is a composite entity of both frequency and severity of hot flashes (The Hot Flash Diary collects the following information for Day 1- Day 7 of each week: Number of mild hot flashes, Number of moderate hot flashes, Number of severe hot flashes, Number of very severe hot flashes). This is a count, so it can range from 0 to infinity.
Time Frame: Baseline up to day 49
Population: Patients who received high-dose oxybutynin, low-dose oxybutynin or placebo and completed the Hot Flash Diary at baseline and Week 7 are included in this analysis. Low-dose and high-dose placebo groups were combined to serve as a control/placebo group to compare with the low-dose and high-dose oxybutynin chloride groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- High-dose Oxybutynin Chloride Group: Patients receive higher dose oxybutynin chloride on days 15-49 in the absence of unacceptable toxicity.
- Placebo Group: Patients receive placebo PO BID on days 8-49 in the absence of unacceptable toxicity.
Arm/Group | High-dose Oxybutynin Chloride Group | Low-dose Oxybutynin Chloride Group | Placebo Group
Number analyzed (Participants) | 31 | 34 | 35
score on a scale | -16.9 (15.6) | -10.6 (7.7) | -5.7 (10.2)
Statistical Analysis 1: Comparison: Low-dose Oxybutynin Chloride Group vs Placebo Group; Test type: Superiority; p = 0.0041, Kruskal-Wallis
Statistical Analysis 2: Comparison: High-dose Oxybutynin Chloride Group vs Placebo Group; Test type: Superiority; p = 0.0001, Kruskal-Wallis

2. Secondary Outcome: Average Change in Hot Flash Score From Week 1 to Week 7 Comparing Low Dose Oxybutynin to Placebo
Description: Average change in Hot Flash Score from Week 1 to Week 7 Comparing Low Dose Oxybutynin to Placebo. The least squares (LS) mean was estimated from a mixed-effects model with repeated measures (MMRM) that included low dose oxybutynin, weeks 1-7, no current aromatase inhibitor, age group 18-49, no tamoxifen, hot flash symptom duration < 9 months, and 4-9 hot flashes/day as fixed effects, and participant and error as random effects. The mean change in Hot Flash Score from Week 1 to Week 7 is reported below for the low-dose oxybutynin and placebo groups.
Time Frame: Baseline up to day 49
Population: Patients who received low-dose oxybutynin or placebo and completed the Hot Flash Diary at baseline and Week 7 are included in this analysis. Low-dose and high-dose placebo groups were combined to serve as a control/placebo group to compare with the low-dose oxybutynin chloride group.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Low-dose Oxybutynin Chloride Group | Placebo Group
Number analyzed (Participants) | 34 | 35
score on a scale | 8.1 (0.63) | 15.6 (0.66)
Statistical Analysis 1: Comparison: Low-dose Oxybutynin Chloride Group vs Placebo Group; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Adjusted for effects specified in outcome measure description

3. Secondary Outcome: Average Change in Hot Flash Score From Week 1 to Week 7 Comparing High Dose Oxybutynin to Placebo
Description: Average change in Hot Flash Score from Week 1 to Week 7 Comparing High Dose Oxybutynin to Placebo. The least squares (LS) mean was estimated from a mixed-effects model with repeated measures (MMRM) that included low dose oxybutynin, weeks 1-7, no current aromatase inhibitor, age group 18-49, no tamoxifen, hot flash symptom duration < 9 months, and 4-9 hot flashes/day as fixed effects, and participant and error as random effects. The mean change in Hot Flash Score from Week 1 to Week 7 is reported below for the high-dose oxybutynin and placebo groups.
Time Frame: Baseline up to day 49
Population: Patients who received higher dose oxybutynin or placebo and completed the Hot Flash Diary at baseline and Week 7 are included in this analysis. Low-dose and high-dose placebo groups were combined to serve as a control/placebo group to compare with the high-dose oxybutynin chloride group.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | High-dose Oxybutynin Chloride Group | Placebo Group
Number analyzed (Participants) | 31 | 35
score on a scale | 9.8 (0.82) | 16.2 (0.82)
Statistical Analysis 1: Comparison: High-dose Oxybutynin Chloride Group vs Placebo Group; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Adjusted for effects specified in outcome measure description

4. Secondary Outcome: Average Change of Severity of Stomach Pain/Cramps Symptoms as Measured by the Symptom Experience Questionnaire From Baseline to Week 7 for Low Dose Oxybutynin vs Placebo and for High Dose Oxybutynin vs Placebo
Description: Average Change of severity of Stomach pain/cramps symptoms as measured by the Symptom Experience Questionnaire From Baseline to Week 7 for Low Dose Oxybutynin vs Placebo and for High Dose Oxybutynin vs Placebo The Symptom Experience Questionnaire stomach pain/cramps item ("Over the past week, have you experienced stomach pain or cramps?") is scored from 0 to 10 with higher values being worse symptoms. So a negative value means the symptom is improving and a positive score means the symptom is getting worse.
Time Frame: Baseline up to day 49
Population: Patients who completed baseline and week 7 Symptom Experience Questionnaire Stomach pain/cramps item were included in this analysis. Low-dose and high-dose placebo groups were combined to serve as a control/placebo group to compare with the low-dose and high-dose oxybutynin chloride groups.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | High-dose Oxybutynin Chloride Group | Low-dose Oxybutynin Chloride Group | Placebo Group
Number analyzed (Participants) | 31 | 35 | 36
change in score on a scale | 0.0 (1.3) | -0.3 (1.5) | -1.4 (2.5)
Statistical Analysis 1: Comparison: Low-dose Oxybutynin Chloride Group vs Placebo Group; Test type: Superiority; p = 0.0174, Kruskal-Wallis
Statistical Analysis 2: Comparison: High-dose Oxybutynin Chloride Group vs Placebo Group; Test type: Superiority; p = 0.0279, Kruskal-Wallis

5. Secondary Outcome: Average Change of Daily Interference (Work) From Baseline to Week 7 as Measured by the Hot Flash-Related Daily Interference Scale (HFRDIS) Comparing Low Dose Oxybutynin vs Placebo and High Dose Oxybutynin vs Placebo
Description: Average Change of daily interference (Work) from baseline to Week 7 as measured by the Hot Flash-Related Daily Interference Scale (HFRDIS) comparing Low dose oxybutynin vs Placebo and High dose oxybutynin vs Placebo. HFRDIS Work item ("Work (work outside the home and housework)") Interference scores run from 0 to 10 with 0 being no interference and 10 being complete interference.
Time Frame: Baseline up to day 49
Population: Patients who completed the Hot Flash-Related Daily Interference Scale (HFRDIS) Work item at baseline and week 7 are included in this analysis. Low-dose and high-dose placebo groups were combined to serve as a control/placebo group to compare with the low-dose and high-dose oxybutynin chloride groups.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | High-dose Oxybutynin Chloride Group | Low-dose Oxybutynin Chloride Group | Placebo Group
Number analyzed (Participants) | 29 | 30 | 32
change in score on a scale | -2.3 (3.4) | -2.9 (3.2) | -0.2 (3.2)
Statistical Analysis 1: Comparison: Low-dose Oxybutynin Chloride Group vs Placebo Group; Test type: Superiority; p = 0.0011, Kruskal-Wallis
Statistical Analysis 2: Comparison: High-dose Oxybutynin Chloride Group vs Placebo Group; Test type: Superiority; p = 0.0025, Kruskal-Wallis

6. Secondary Outcome: Toxicity, Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (v4)
Description: The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns within patient groups. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Up to 7 weeks
Population: Patients who received at least one cycle of treatment and were assessed for adverse events were included in this analysis. Low-dose and high-dose placebo groups were combined to serve as a control/placebo group to compare with the low-dose and high-dose oxybutynin chloride groups.
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose Oxybutynin Chloride Group | Low-dose Oxybutynin Chloride Group | Placebo Group
Number analyzed (Participants) | 45 | 48 | 44
Participants
  grade 3 | 1 | 1 | 0
  grades 4/5 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the end of each cycle for patients randomized to the treatment arm; Up to 7 weeks
Description: All graded AEs are reported for patients who completed at least 1 cycle of tx & AEs were assessed. The high dose and low dose placebo arms are combined for adverse event reporting. Because patients on these two arms are all taking placebo (and nothing else), there is no reason for adverse events to be different on these two placebo arms. This is consistent with the analysis of the primary endpoint, where each Oxybutynin arm was compared with the combined placebo arms.
Groups:
- Placebo Group: Patients receive placebo regardless of dose level in the absence of unacceptable toxicity.
Arm/Group | High-dose Oxybutynin Chloride Group | Low-dose Oxybutynin Chloride Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/48 | 0/44
Serious Adverse Events (participants affected / at risk) | 2/46 | 0/48 | 0/44
Other Adverse Events (participants affected / at risk) | 19/46 | 13/48 | 8/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-dose Oxybutynin Chloride Group (N=46) | Low-dose Oxybutynin Chloride Group (N=48) | Placebo Group (N=44)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-dose Oxybutynin Chloride Group (N=46) | Low-dose Oxybutynin Chloride Group (N=48) | Placebo Group (N=44)
Blurred vision (Eye disorders) | 3 (3) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 3 (8) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (8)
Dry mouth (Gastrointestinal disorders) | 14 (41) | 10 (26) | 3 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4) | 0 (0)
Concentration impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 3 (8) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (5) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (5) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT02961790/Prot_SAP_000.pdf